CLINICAL TRIAL: NCT02206399
Title: Non-Invasive Hemoglobin Multi-Center Observational Study
Brief Title: Non-Invasive Hemoglobin Study
Status: Completed | Type: Observational
Sponsor: Convergence Biometrics (Industry)
Collaborators: DRMiller Engineering (Unknown)
Responsible Party: Sponsor
Other Study IDs: BLS-1
Record Dates: First submitted 2014-07-25; First posted 2014-08-01 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The investigators clinical trials will be for a medical device that is non-invasive in nature. The investigators will be studying whether their non-invasive medical device gets data that is as good as, or better than, an FDA previously approved, blood analysis device. There is no study hypothesis for this study.

ELIGIBILITY:
Inclusion criteria for this study are:

1. Subject is capable of giving informed consent.
2. Subject has an anatomically intact digit capable of having a capillary sample taken and of being placed in the POCT device.

Exclusion criteria for this study are:

1. Age less than 18 years at time of research
2. Subject lacks the digits to place in the POCT device
3. Subject displays symptoms or has a history of Raynaud's disease
4. Subject has a neurological disorder resulting in an inability to hold the index finger steady for 20 sec.
5. Subject has a history of long term continuous decreased perfusion to either hand (>30 days).
6. Subject has had surgery within the last 2 weeks on finger or hand that he wishes to use in the study
7. Subject's same day participation in this study
8. Capillary sample volume is not adequate to complete testing on the comparative device.
9. Cold agglutinin disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Whole Blood Donation Center Donors sample
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Hemoglobin in Blood At Time of Test | Up to 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Anne Igbokwe, MD, Principal Investigator — BloodSource; Chris Gresens, MD, Principal Investigator — BloodSource
Locations (1):
- BloodSource, Sacramento, California, United States